CLINICAL TRIAL: NCT04300387
Title: Biomarker and Multidisciplinary Predialysis Education in Chronic Kidney Disease Patients
Brief Title: Chronic Kidney Disease at Northeast Taiwan: Biomarker and Multidisciplinary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, I Wen Wu, MD, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IWW-0005
Record Dates: First submitted 2016-09-30; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Chronic Kidney Disease
Keywords: risk factors; omics; multidisciplinary care
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Patient Care Team

ARMS (2):
- customary care (No Intervention): customary care for CKD
- multidisciplinary care (Active Comparator): multidisciplinary team care for CKD
  Interventions: Behavioral: multidisciplinary care

INTERVENTIONS:
Behavioral: multidisciplinary care — multidisciplinary CKD care involving case management nurse, dietitian, social worker, pharmacists.
  Arms: multidisciplinary care

SUMMARY:
CKD is a global endemic disease with increased comorbidities and mortality. The prevalence and the incidence of the end-stage renal disease (ESRD) are extremely high in Taiwan. Early diagnosis of disease and proper management remain challenging. The aims of this study are:

1. Explore risk factors associated with CKD
2. Establish multidisciplinary care model for CKD patients
3. Development cost-effective clinical care pathway for CKD
4. Provide bio-specimen repository for future study

DETAILED DESCRIPTION:
CKD is a global endemic disease with increased comorbidities and mortality. The prevalence and the incidence of the end-stage renal disease (ESRD) are extremely high in Taiwan. Early diagnosis of disease and proper management remain challenging. The aims of this study are:

1. Explore risk factors associated with CKD: demographic, social and genetics factors
2. Establish multidisciplinary care model for CKD patients
3. Development cost-effective clinical care pathway for CKD
4. Provide bio-specimen repository for future study: serum, PBMC, urine and stool

ELIGIBILITY:
Inclusion Criteria:

* Subjects visiting outpatient clinics of nephrology of Chang Gung Memorial Hospital

Exclusion Criteria:

* Patient receiving dialysis or transplantation
* Unwilling to participate

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2011-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
percentage (%) | through study completion, every 1 year
  percentage of patients with new CKD, starting dialysis treatments, cardiovascular event or mortality
difference of US dollars | through study completion, every 1 year
  differences of US dollars of medical care (out patients and inpatients service fees) between groups

SECONDARY OUTCOMES:
fold changes of proteins | through study completion, every 1 year
  change of levels between groups
fold changes of microRNA | through study completion, every 1 year
  change of levels between groups

OTHER OUTCOMES:
change of taxonomic units abundance of specific microbiota | through study completion, every 1 year
  change of levels between groups
changes of metabolites | through study completion, every 1 year
  change of levels between groups

CONTACTS AND LOCATIONS:
Overall Officials: I-Wen Wu, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Keelung, Taiwan

REFERENCES:
- [Result] Wu IW, Wang SY, Hsu KH, Lee CC, Sun CY, Tsai CJ, Wu MS. Multidisciplinary predialysis education decreases the incidence of dialysis and reduces mortality--a controlled cohort study based on the NKF/DOQI guidelines. Nephrol Dial Transplant. 2009 Nov;24(11):3426-33. doi: 10.1093/ndt/gfp259. Epub 2009 Jun 2. PMID 19491379
- [Result] Chen SH, Tsai YF, Sun CY, Wu IW, Lee CC, Wu MS. The impact of self-management support on the progression of chronic kidney disease--a prospective randomized controlled trial. Nephrol Dial Transplant. 2011 Nov;26(11):3560-6. doi: 10.1093/ndt/gfr047. Epub 2011 Mar 17. PMID 21414969